CLINICAL TRIAL: NCT01005420
Title: The Effect of Anthocyanins in the Form of Blueberry Powder on Enhancing Insulin Sensitivity in Insulin Resistant and Obese Humans
Brief Title: The Effect of Blueberries on Enhancing Insulin Sensitivity in Humans: A Pilot Study
Acronym: BLUEBERRY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled and was closed in IRB February 24, 2015
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PBRC 27030
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2022-09

CONDITIONS: Insulin Sensitivity
Keywords: Insulin Sensitivity; Pre-diabetes; Diabetes; Blueberries; Anthocyanins
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Powder (Experimental): A blueberry smoothie will be consumed at the breakfast and dinner meals.
  Nutritional Value:(based on one 16oz smoothie and subjects had to consume two a day)
  * 206.4 Kcals
  * 40.3 g Carbohydrate
  * 11.5 g Protein
  * 0.08 g Fat
  * 0.05 g Sat fat
  * 4.2 g Fiber
  Ingredients:
  * 245.0 g Dannon Light & Fit yogurt
  * 105 .0 g Skim milk
  * 22.5 g Freeze-dried blueberry powder
  * 5.0 g Imitation vanilla flavor
  * 1.0 g Splenda
  * 16 oz plastic cup with lid
  * Smoothie total weight - 378.5 g
  Interventions: Dietary Supplement: Blueberry Powder
- Placebo (Placebo Comparator): A placebo smoothie will be consumed at the breakfast and dinner meals.
  Nutritional Value:(based on one 16oz smoothie and subjects had to consume two a day)
  * 201.3 Kcals
  * 40.3 g Carbohydrate
  * 10.7 g Protein
  * 0.08 g Fat
  * 0.05 g Sat fat
  * 4.3 g Fiber
  Ingredients:
  * 245.0 g Dannon Light & Fit yogurt
  * 105 .0 g Skim milk
  * 5.0 g Benefiber
  * 12.0 g Sugar
  * 4.0 g Artificial blueberry flavor(liquid & powder)
  * 1.5 g Red food color
  * 0.7 g Blue food color
  * 16 oz plastic cup with lid
  * Smoothie total weight - 373.2 g
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberry Powder — The blueberry and placebo groups will be randomized to receive 45g of blueberry powder or control per day. Blueberry powder will be given as a smoothie to be consumed at the breakfast and dinner meals and an identical smoothie will be given as a control. The smoothies will be prepared in the metabolic kitchen and a week supply of frozen smoothies will be given to participants. Both the blueberry powder and control smoothie contain comparable energy and macronutrients.
  Arms: Blueberry Powder
Dietary Supplement: Placebo — The blueberry and placebo groups will be randomized to receive 45g of blueberry powder or control per day. Blueberry powder will be given as a smoothie to be consumed at the breakfast and dinner meals and an identical smoothie will be given as a control. The smoothies will be prepared in the metabolic kitchen and a week supply of frozen smoothies will be given to participants. Both the blueberry powder and control smoothie contain comparable energy and macronutrients.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of blueberry powder on insulin sensitivity in obese, non-diabetic, and insulin resistant subjects. The investigators hypothesized that supplementation with blueberry powder will result in an increase in insulin sensitivity in obese subjects with insulin resistance.

DETAILED DESCRIPTION:
Insulin resistance is a key pathophysiologic feature of the "metabolic syndrome" and is strongly associated with co-existing cardiovascular risk factors and accelerated atherosclerosis. Due to the clinical consequences associated with insulin resistance in subjects with metabolic syndrome and type 2 diabetes, clinical regimens directed at increasing insulin sensitivity in vivo remain one of the most desirable goals of treatment. Although it is well established that lifestyle modification can improve insulin resistance and effectively improve many of the risk factors associated with the metabolic syndrome, the success of maintaining lifestyle changes in humans over a chronic period is poor. Therefore, strategies to improve insulin resistance by pharmacological means have represented the traditional approach for clinical medicine. However, because of the widespread use of dietary supplements by the general public, nutritional supplementation with the use of botanical extracts that effectively increase insulin sensitivity represent a very attractive and novel approach.

Unfortunately, considerable controversy exists regarding the effect of botanical supplements on the metabolic syndrome in large part because efficacy data for many of the supplements used for this purpose consists of only uncontrolled studies and anecdotal reports. As such, there is a paucity of data in humans in regard to the effect of botanicals to improve measures of insulin action in vivo or on cellular aspects of insulin action. However, several lines of evidence in both in vitro and in vivo models suggest that botanicals may modulate intracellular pathways of glucose metabolism. Specifically, preclinical data with use of extracts from grapes and blueberries suggest that components of these botanical mixtures, e.g. anthocyanins and resveratrol, may play a role in enhancing cellular pathways of insulin action. On a clinical level, if cellular pathways of insulin action are enhanced, e.g. PI-3 kinase activity, this should be associated with an increase in whole body glucose disposal as reflected in measures assessing insulin sensitivity. However, there is limited experience in human studies for which insulin sensitivity has been assessed with use of "gold standard" techniques assessing in vivo insulin action. Therefore, this project's overall objective is to examine the role of a specific botanical (i.e., blueberry powder) on insulin action in vivo with use of hyperinsulinemic-euglycemic clamps. This pilot trial is designed to evaluate a fixed consumption of blueberry powder and to provide data of the effect so that a larger, more comprehensive study can be planned. To accomplish our goal, we will conduct a randomized, placebo-controlled pilot clinical study with blueberry powder designed to assess insulin sensitivity in subjects who are obese and insulin resistant. We hypothesize that blueberry powder will be effective, when compared to placebo, to increase insulin action in vivo. If so, this pilot trial will provide the necessary background to progress to studies in subjects with Type 2 diabetes. An increase in insulin sensitivity in patients with Type 2 diabetes will be expected to markedly reduce glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 20 years of age.
* Subjects not currently treated with diabetes medication.
* Subjects with fasting blood glucose at time of screening is ≤ 110 mg/dL.
* Subjects with a Body Mass Index (BMI) ≥ 32 and ≤ 45.
* Written Informed Consent obtained PRIOR to performing any screening tests or study procedures.
* Subjects who have glucose disposal rate ≤ 650 mg/min assessed clinically at visit 4

Exclusion Criteria:

* Subjects with a prior history of Type 2 diabetes.
* Women who are pregnant or who are lactating.
* Women of childbearing potential who are not using an effective method of birth control, condoms with spermicidal gel or foam, contraceptive patch, are not surgically sterilized, or not at least 2 years postmenopausal.
* Subjects who have type 1 diabetes.
* Subjects who are currently on thiazolidinediones (rosiglitazone or pioglitazone) or who have taken these agents in the previous 12 weeks.
* Subjects who are on concomitant therapy with glucocorticoids (except topical or inhalant glucocorticoids). Other medications that have an effect on glucose homeostasis (i.e. ACE inhibitors) are acceptable if they have been administered in a stable dosage during the preceding 6 months and dosage will continue unchanged during the study.
* Subjects with a history or evidence of significant gastrointestinal dysfunction.
* Subjects who have chronic use of laxatives or cathartics. The use of stool softeners is acceptable. Use of bulking agents, if required, should remain constant.
* Subjects who are taking concomitant therapy with medications known to be nephrotoxic, such as aminoglycosides, methicillin, and cyclosporin.
* Subjects who have evidence of clinically significant renal dysfunction or disease, e.g. serum creatinine >1.5 mg/dL in males and >1.4 mg/dL in females and/or BUN >50 mg/dL, proteinuria of >1 gram/day or 4+ proteinuria on dipstick urinalysis.
* Subjects with clinically significant cardiovascular dysfunction and/or history (within the preceding 6 months) of significant cardiovascular dysfunction, e.g., congestive heart failure or serious arrhythmia, myocardial infarction, cardiac surgery; transient ischemic attacks or cerebrovascular accident during the preceding six months; diagnosis of symptomatic autonomic neuropathy with a history of orthostatic hypertension, syncope, or hypertension with a systolic blood pressure of ≥180 mm Hg and diastolic blood pressure ≥110 mm Hg at the time of screening visit.
* Subjects who have evidence within the preceding 6 months of hepatic disease or dysfunction, e.g. AST, ALT, alkaline phosphatase or total bilirubin twice the upper limit of normal; hepatitis; jaundice; cirrhosis.
* Subjects with clinically significant pulmonary, neurologic, hematologic, immunologic, neoplastic or metabolic disease.
* Subjects with evidence or recurrence of malignancy within the past five years, other than excised basal cell carcinoma.
* Subjects for whom surgery is anticipated during the study period.
* Subjects with an history of substance abuse or alcoholism within the past 5 years, or significant psychiatric disorder that would interfere with the subject's ability to complete the study.
* Subjects who have donated blood during the month prior to study entry or planned during the study.
* Subjects who have participated in other studies using an investigational drug during the preceding 3 months.
* Subjects who are current smokers or have smoked within the previous 6 months. No smoking will be allowed during the study.
* Subjects who are allergic to blueberries.
* Subjects who are lactose intolerant.
* Subjects who consume and drink daily servings of berries (i.e., blueberries, strawberries, bilberries, cranberries, elderberries, and raspberries), grapes, fruit juices that contain berries and grapes, and wine more than 3 times per week.
* Subjects that have had a fluctuation in body weight >5% in the preceding 2 months.
* Subjects who are taking prescription or over the counter medication or supplements for desired weight loss.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | before intervention (Week 0) and 6 weeks after intervention started

SECONDARY OUTCOMES:
Cognitive Performance | screening and 5 weeks after intevention started

CONTACTS AND LOCATIONS:
Overall Officials: William T Cefalu, MD, Principal Investigator — Pennington Biomedical Research Center; April Stull, Ph.D., Study Director — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Stull AJ, Cash KC, Johnson WD, Champagne CM, Cefalu WT. Bioactives in blueberries improve insulin sensitivity in obese, insulin-resistant men and women. J Nutr. 2010 Oct;140(10):1764-8. doi: 10.3945/jn.110.125336. Epub 2010 Aug 19. PMID 20724487